CLINICAL TRIAL: NCT01964586
Title: Phase 4 Study of Comparison of Preincisional Infiltrated Dexmedetomidine and Lidocaine Plus Adrenaline for Surgical Conditions and Postoperative Analgesic Consumption in Nasal Sephoplasty Surgery.
Brief Title: Comparison of Preincisional Infiltrated Dexmedetomidine and Lidocaine Plus Adrenaline for Nasal Sephoplasty Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Adnan Bayram, Asst Prof, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2013/167
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Surgery; Pain
Keywords: Septoplasty, Dexmedetomidine, Surgical Conditions
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine plus Adrenaline (Active Comparator): Lidocaine and adrenaline diluted to 10 ml with normal salin and infiltrated to both side of the nasal septum before 10 minutes from the surgery.
  Interventions: Drug: Lidocaine; Drug: Adrenaline
- Dexmedetomidine (Active Comparator): 2 mcg/kg dexmedetomidine diluted to 10 ml with normal salin and infiltrated to both side of the nasal septum before 10 minutes the surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 2 mcg/kg dexmedetomidine was administered 10 minutes before the surgery by infiltration to the both side of the nasal septum.
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Lidocaine — 10 ml 2% lidocaine was administered 10 minutes before the surgery by infiltration to the both side of the nasal septum.
  Other Names: Jetokain %2
  Arms: Lidocaine plus Adrenaline
Drug: Adrenaline — 12.5 mcg/ml 10 ml adrenaline was administered 10 minutes before the surgery by infiltration to the both side of the nasal septum.
  Other Names: Adrenalin; Epinefrin
  Arms: Lidocaine plus Adrenaline

SUMMARY:
It is very important to decrease the bleeding during nasal septoplasty in order to increase the visibility of the surgical site. Our primary goal was to investigate the effects of dexmedetomidine and lidocaine plus adrenaline on visibility of surgical site and postoperative analgesic consumption.

DETAILED DESCRIPTION:
Nasal septoplasty is a surgery procedure which needs to have decrease the bleeding during the surgery for the visibility of surgical site.And postoperative pain is very usual after the surgery, so an effective postoperative analgesia procedure reduces the complications and helps to be discharged earlier from the hospital. An alpha 2 agonist Dexmedetomidine has an analgesic effect and vasoconstructive effect on the periferal blood vessels. Our hypothesis was dexmedetomidine makes a better surgecal conditions during the surgery and reduce the postoperative analgesic consumption. We administered the infiltrated dexmedetomidine or lidocaine plus adrenaline to the both side of the nasal septum 10 minutes before the surgery. Bleeding scores (Fromm and Boezaart Bleeding Scores) were recorded during the surgery. And postoperative analgesic consumptions were recorded in first 24 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for the nasal septoplasty surgery
* ASA 1-2 patients
* 18-60 yo patients

Exclusion Criteria:

* Pregnant patients
* ASA 3-4 patients
* Under 18 yo childrens

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
surgical conditions | during the surgery
  Bleeding scores were recorded during the surgery

SECONDARY OUTCOMES:
Analgesic Consumption | Up to 24 hours
  Analgesic consumption were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Bayram, MD, Principal Investigator — TC Erciyes University